CLINICAL TRIAL: NCT04640584
Title: A Prospective Registry of Patients Fitted With a Microprocessor-controlled Knee Ankle Foot Orthosis
Brief Title: C-Brace Prospective Registry
Status: Recruiting | Type: Observational
Sponsor: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PD-PS00120018A-001
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pareses; Lower Extremity
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: C-Brace — The C-Brace consists of individually fabricated thigh, calf and foot components. An ankle joint, unilateral or bilateral fitting, or an individual spring element connects the foot and calf components. The sensor system continuously measures the flexion of the knee joint and its angular acceleration. This allows the C-Brace to detect the user's current walking phase, so it can regulate the hydraulic resistances as well as control the flexion and extension of the knee joint.
  Other Names: Microprocessor-controlled Stance and Swing Orthosis (MP-SSCO)

SUMMARY:
To gather prospective safety and effectiveness data for the C-Brace System following the standard of care.

DETAILED DESCRIPTION:
The purpose of the C-Brace Prospective Registry is to gather prospective baseline and follow-up data to characterize the safety and effectiveness of the C Brace. Patients casted for C-Brace fitting and willing to provide informed consent at participating clinics will be enrolled in the registry. All patients will be followed in accordance with the standard of care for a C-Brace, which will include, at a minimum, baseline evaluation, fitting, patient training/therapy sessions, follow-up at 6 months, 12 months, 24 months and 36 months after the definitive fitting of the C-Brace.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been evaluated and successfully tested with the Trial Tool, and has been casted for a C-Brace.
* Patient is able to communicate, provide feedback, understand and follow instructions during the course of the registry.
* Patient is willing to provide informed consent.

Exclusion Criteria:

* Patient is geographically inaccessible to comply and participate in the registry.
* Patient has not been casted for a C-Brace fitting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As the purpose of the C-Brace Registry is to characterize safety and effectiveness data in a real-world setting, the inclusion and exclusion criteria are deliberately written as open as possible to allow all patients casted for a C-Brace fitting to be included as subjects in the registry. The indications and contraindications for the C-Brace are provided in the Instructions for Use and are based on clinical presentation, not on etiology. Clinical presentations will involve lower limb paresis that may be due to a variety of etiologies, including incomplete paraplegia, post-polio syndrome, peripheral neuropathy, traumatic brain injury and muscular sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy: Timed Walk Test | Change in walking speed with the C-Brace measured either by a 25-ft or 10-m walk test compared to baseline measurements when assessed 12 months after initial fitting
  The Timed Walk test is used to measure gait speed on either a 25-foot or 10-meter straight course timed using the middle 10 feet or 6 meters, respectively. Three trials are performed and the average of the three used. Patients are allowed the use of assistive device (such as a cane, crutches or walker) that they normally use for in home or community ambulation.
Primary Efficacy: Timed Up and Go (TUG) Test | Changes in mobility, balance, risk of falling, and walking ability as measured by TUG test with the C-Brace system compared to baseline when assessed 12 months after the initial fitting.
  Originally designed to test mobility skills in the elderly, the TUG is a validated test for quantifying functional mobility and risk of falling. In the TUG Test, patients are asked to stand up from a chair, walk ten feet, turn and return to the chair, and then sit on the chair. For centers routinely using the TUG as a part of their standard of care, this data (time to complete in seconds) will be collected at baseline and follow-up visits when available. Predictive results from the test are as follows: <10s, Freely mobile; < 20s, Mostly independent; 20-29s, Variable mobility.
Primary Efficacy: Activities-specific Balance Confidence (ABC) | Changes in perceived balance confidence as assessed by the ABC score with the C-Brace system compared to baseline when assessed 12 months after the initial fitting.
  Assessment of patient-perceived balance confidence for 16 activities of daily living. For each activity, subjects rate their level of confidence in doing the activity without losing their balance or becoming unsteady on a scale from 0% to 100%, with 100% being the highest level of confidence. The total score for the ABC scale is an average of all activity scores.
Primary Safety: Frequency and severity of falling | Changes in numbers of device-related adverse events experienced by C Brace users by frequency and severity compared to baseline measurement when assessed 12 months after the initial fitting
  The number and percentage of patients who experience one or more adverse events during their participation in the registry will be computed along with the exact 95% binomial confidence interval. The number and percentage of subjects who experience a serious adverse event will also be tabulated along with the exact 95% binomial confidence interval. Events will also be categorized and the number of events and number of patients for each category will be presented. In addition, a complete listing of adverse events along with their relationship to the device, severity, seriousness and outcome will be constructed.

SECONDARY OUTCOMES:
Patient Specific Functional Scale (PSFS) | Changes in patient-centered activities and in the defined activity performance with C-Brace by the PSFS compared to baseline when assessed 12 months after the initial fitting.
  The PSFS is a self-report measure aimed at identifying functional status limitations that are most relevant to individual patients.The PSFS is a reliable, valid, and efficient measure for detecting clinical change in persons with low back pain and knee dysfunction. Patients will be asked to identify three to five activities that they are having difficulty or are unable to perform because of their injury/condition. For the specified activities, patients will then be asked to rate their ability to perform each activity at that time (0-10 numerical scale) with '0' being unable to perform the activity, and '10' being able to perform the activity at the same level as they could prior to the injury/condition. There is no total score for this measure.
Activity Tracker | Changes of C-Brace utilization at 12 months compared to baseline measurement estimated by the activity tracker
  On the day the patient is casted for the C-Brace the patient's current orthosis will be affixed with an activity monitor to record the number of steps the patient takes with the orthosis. The patient will be sent home with a prepaid envelope and be instructed to mail back the activity monitor 16 days later, in order to capture 14 whole days of step count data. The step counts will be downloaded from the device the day the activity monitor is returned to the Investigator. The C-Brace will also be affixed with the same activity monitor following the same process for when the activity monitor was attached to the previous orthosis.
Berg Balance Scale (BBS) | Changes in static and dynamic balance abilities as measured by the BBS compared to baseline when assessed 12 months after initial fitting with C-Brace.
  The BBS is a 14-item scale designed to measure static and dynamic balance in adults in a clinical setting. The range in score for the BBS is 0 to 56, with higher scores indicating better balance. Points for each item are deducted if the time or distance requirements are not met, the patient's performance requires supervision, or the patient requires assistance from support or examiner. The points reached in each item were summed up to the total score.

OTHER OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Reduction in joint, lower back, and limb pain as measured by the NPRS compared to baseline when assessed 12 months after the initial fitting with C-Brace.
  The NPRS is a valid and reliable measure of pain that may be used across all musculoskeletal injuries/conditions and complements the Patient Specific Functional Scale (PSFS). The patient will be asked to rate the pain of their joints, foot, lower back, and if they are using an assistive device any additional affected limbs on average over the last 24 hours on a scale 1-10, with '1' being 'very mild' and '10' being the 'unimaginable unspeakable'. There is no total score for the NPRS.
Manual Muscle Test | Changes in muscle strength and function as measured by the Manual Muscle Test (MMT) compared to baseline when assessed 12 months after initial fitting.
  The Manual Muscle Test is using a grading system of 0-5 in muscles of the lower body (hip, knee, ankle), 0 indicating none muscle strength at all, 5 means normal. In addition, assessments for range of motion, contractures, and alignment in the lower limb will all be recorded.There is no total score for these assessments
EQ-5D-5L | Changes in health-related quality of life as assessed by the EQ-5D-5L with the C-Brace system compared to baseline when assessed 12 months after the initial fitting.
  Measure of health status composed of 5 dimensions: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, anxiety and depression. Each dimension is rated on a 5-point scale indicating the level of perceived problems for each dimension (level 1 indicating no problems and level 5 indicating extreme problems). Each health state can potentially be assigned a summary index score based on societal preference weights for the health state. These weights, sometimes referred to as 'utilities', are often used to compute QALYs for use in health economic analyses. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
PROMIS Pain Interference - Short Form 6a | Reduction in the consequences of pain as measured by the PROMIS Pain Interference Short form 6a compared to baseline when assessed at 12 months after the initial fitting.
  PROMIS item banks and their short forms are a reliable and precise measurements of patient reported outcome measures. For this registry the Pain Interference - Short Form 6a has been chosen for use by the patient. The patient will be asked six questions related to how pain may have interfered with certain activities in the last 7 days, and rate them on a 1-5 scale, with '1' being 'not at all' and '5' being 'very much.' To find the total raw score for the short form, the values of the responses are summed. The raw score is then converted to a T-Score. A higher PROMIS T-score represents more of the concept being measured.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Braatz, Prof., Principal Investigator — Private University of Applied Sciences
Locations (76):
- United States (70):
  - Jonesboro P&O x Ottobock.care, Harrison, Arkansas
  - Jonesboro P&O x Ottobock.care, Rogers, Arkansas
  - Bionics Orthotics & Prosthetics, San Diego, California
  - ABI P&O, San Diego, California
  - West Coast Brace & Limb - Palm Harbor, Palm Harbor, Florida
  - Hanger - Sarasota, Sarasota, Florida
  - West Coast Brace & Limb - Tampa, Tampa, Florida
  - ProCare Prosthetics x Ottobock.care, Buford, Georgia
  - ProCare x Ottobock.care, Conyers, Georgia
  - Scheck & Siress: A Hanger Clinic Company, Chicago, Illinois
  - P&O Care x Ottobock.care, Fairview Heights, Illinois
  - Kenney Orthopedics - Evansville, Evansville, Indiana
  - Prevail Prosthetics & Orthotics, Fort Wayne, Indiana
  - Bionic Prosthetics & Orthotics, Merrillville, Indiana
  - Kenney Orthopedics - Danville, Danville, Kentucky
  - Kenney Orthopedics - Lexington, Lexington, Kentucky
  - Ability x Ottobock.care, Frederick, Maryland
  - Dankmeyer, Linthicum, Maryland
  - Medical Center Orthotics & Prosthetics, Silver Spring, Maryland
  - Cornell Orthotics & Prosthetics, Beverly, Massachusetts
  - Wright & Filippis x Ottobock.care, Clinton Township, Michigan
  - Wright & Filippis x Ottobock.care, Farmington Hills, Michigan
  - Wright & Filippis x Ottobock.care, Flint, Michigan
  - Wright & Filippis x Ottobock.care, Lansing, Michigan
  - Wright & Filippis x Ottobock.care, Lapeer, Michigan
  - Wright & Filippis x Ottobock.care, Livonia, Michigan
  - Wright & Filippis x Ottobock.care, Madison Heights, Michigan
  - Limb Lab, Rochester, Minnesota
  - P&O Care x Ottobock.care, St Louis, Missouri
  - Limb Lab, Omaha, Nebraska
  - AlliedOP, Fair Lawn, New Jersey
  - AlliedOP, Mount Laurel, New Jersey
  - MedEast Post-op & Surgical, Mount Laurel, New Jersey
  - Body in Motion, Toms River, New Jersey
  - Raymond G. Murphy VA, Albuquerque, New Mexico
  - Orthocraft Inc. - 3856 Flatlands Ave, Brooklyn, New York
  - VA NY Harbor, Manhattan, New York
  - Prosthetics in Motion, New York, New York
  - Reliable P&O, Jacksonville, North Carolina
  - Bionic Prosthetics & Orthotics, Lenoir, North Carolina
  - O&P of Pinehurst, Pinehurst, North Carolina
  - Atlantic Prosthetic Services, Wilmington, North Carolina
  - Yanke Bionics - W Exchange St, Akron, Ohio
  - Western Reserve O&P, Austintown, Ohio
  - Ability P&O x Ottobock.care, Exton, Pennsylvania
  - Titleman Orthopedic, Philadelphia, Pennsylvania
  - elizur Corporation, Pittsburgh, Pennsylvania
  - Ability x Ottobock.care, Wyomissing, Pennsylvania
  - Ability x Ottobock.care, York, Pennsylvania
  - South County Artificial Limb and Brace, Wakefield, Rhode Island
  - Carolina Ottobock.care, Spartanburg, South Carolina
  - Excel P&O, Kingsport, Tennessee
  - Restorative Health Services, Murfreesboro, Tennessee
  - Ottobock.care, Austin, Texas
  - New Life, Conroe, Texas
  - Scott Sabolich Prosthetics & Research x Ottobock.care, Dallas, Texas
  - Baker O&P, Fort Worth, Texas
  - Hanger Clinic - Houston, Houston, Texas
  - Michael E. DeBakey VA, Houston, Texas
  - TIRR Research Center, Houston, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Freedom P & O - 356 E 600 S, St. George, Utah
  - Hunter Holmes McGuire VA, Richmond, Virginia
  - VA O&P, Roanoke, Virginia
  - Cornerstone P&O, Everett, Washington
  - Cascade Prosthetics & Orthotics, Ferndale, Washington
  - Hanger Clinic - Renton, Renton, Washington
  - Pacific Medical, Richland, Washington
  - Thompson's O&P, Spokane, Washington
  - Bionic Prosthetics & Orthotics, Green Bay, Wisconsin
- Neuromuscular-orthotics.com.au, Clayton, Victoria, Australia
- Germany (4):
  - Pohlig BmbH, Traunstein, Bavaria
  - Ottobock Göttingen, Göttingen, Deutschland
  - John+Bamberg GmbH & Co. KG, Hanover, Lower Saxony
  - Katholisches Klinikum Koblenz-Montabaur, Koblenz, Rhineland-Palatinate
- Hyogo Rehabilitation Hospital, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lundstrom RL, Klenow TD, Morris A, Pobatschnig B, Hibler KD, Kannenberg AH. The C-Brace(R) microprocessor controlled stance and swing orthosis improves safety, mobility, and quality of life at one year: Interim results from a prospective registry. J Rehabil Assist Technol Eng. 2024 Aug 9;11:20556683241269539. doi: 10.1177/20556683241269539. eCollection 2024 Jan-Dec. PMID 39132469